CLINICAL TRIAL: NCT07350252
Title: Postoperative Analgesia in Patients Undergoing Knee Replacement Surgery - a Study Comparing Intraoperative Local Infiltration Analgesia Only With Ultrasound-guided Nerve Blocks Added to Intraoperative Local Infiltration Analgesia, a Randomized Clinical Trial
Brief Title: Combination of Nerve Blocks and Local Infiltration Analgesia in Knee Arthroplasty
Acronym: BALIA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Greta and Johan Kock Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-06626-01
Record Dates: First submitted 2025-12-22; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Osteo Arthritis of the Knee
Keywords: Treatment
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial Number of Arms: 2 parallel arms Allocation Ratio: 1:1 randomization using computer-generated sequence Blinding: Outcome assessor blinded; staff registering NRS pain scores and opioid consumption are blinded to group allocation. No sham block is used in the control group
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Outcome assessor blinded; staff registering NRS pain scores and opioid consumption are blinded to group allocation. No sham block is used in the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm-Nerve blocks in addition to Local Infiltration Analgesia (Active Comparator): Ultrasound guided nerve blocks are administered preoperatively in addition to the Local Infiltration Analgesia administered during surgery.
  Nerve blocks used:
  1. Nerve to Vastus Medialis (NVM) block:
     Injection: 5 ml ropivacaine 5% with clonidine 1.875 micrograms per ml
  2. Saphenous Nerve (SN) block:
     Injection: 10 ml ropivacaine 0.5% with clonidine 1.875 micrograms per ml
  3. Anterior Femoral Cutaneous Nerve (AFCN) Block:
  AFCN divides into multiple branches at the level of the femoral triangle Injection: 1 ml ropivacaine 5% with clonidine 1.875 micrograms per ml per branch
  Local Infiltration Analgesia (LIA):
  150 ml ropivacaine 2 mg/ml with 0.5 mg adrenaline is infiltrated periarticular around the knee capsule, collateral ligaments, under the patella, and subcutaneously
  Interventions: Drug: Ropivacain 5 mg/ml + Clonidine
- Control arm - Local Infiltration Analgesia only (No Intervention): No ultrasound guided nerve blocks are administered. Local Infiltration Analgesia (LIA) is the same as in the- intervention arm:
  150 ml ropivacaine 2 mg/ml with 0.5 mg adrenaline is infiltrated periarticular around the knee capsule, collateral ligaments, under the patella, and subcutaneously

INTERVENTIONS:
Drug: Ropivacain 5 mg/ml + Clonidine — Drug used in the block
  Arms: Intervention Arm-Nerve blocks in addition to Local Infiltration Analgesia

SUMMARY:
The aim of this clinical randomized trial is to compare local infiltration analgesia (LIA) alone versus the combination of LIA with saphenous nerve (SN) block, block of the nerve to vastus medialis (NVM), and anterior femoral cutaneous nerve (AFCN) block in participants undergoing total knee arthroplasty (TKA). The primary outcome is pain intensity, measured using the Numerical Rating Scale (NRS) at multiple time points after surgery. Secondary outcomes include opioid consumption, time to mobilization, postoperative nausea and vomiting, length of hospital stay, neurological complications and differences in opioid consumption and NRS pain scores between general and spinal anesthesia.

DETAILED DESCRIPTION:
Scientific Rationale and Background Total Knee Arthroplasty (TKA) requires effective perioperative pain management. Traditionally, Local Infiltration Analgesia (LIA)has been the standard method, sometimes combined with femoral nerve block. However, femoral nerve block impairs quadriceps motor function, making early mobilization-critical for postoperative rehabilitation-difficult for participants.

Recent advances have introduced purely sensory nerve block techniques that preserve motor function. The knee joint innervation is complex and involves multiple neural pathways. The Saphenous Nerve (SN), Nervus Vastus Medialis (NVM), and the Anterior Femoral Cutaneous Nerve (AFCN) are all branches of the femoral nerve that provide sensory innervation to the knee without contributing to motor control of the quadriceps. The adductor canal contains the SN and NVM, which are primarily sensory nerves. The AFCN travels superficially in the femoral triangle and innervates the skin of the anterior and medial thigh.

Studies have shown that adductor canal block (targeting SN and NVM) combined with LIA provides comparable pain relief to femoral nerve block without motor impairment. Additionally, the AFCN contributes to sensory innervation of the anterolateral and anteromedial aspects of the knee joint. Our hypothesis is that combining these three sensory blocks (SN, NVM, and AFCN) with LIA may provide superior pain control and reduced opioid consumption compared to LIA alone, while preserving motor function necessary for early mobilization.

Primary Research Questions

1. Does the combination of the SN block, the NVM block of and the AFCN block togheter with LIA provide better postoperative pain control compared to LIA alone?
2. Does the above combination reduce total postoperative opioid consumption? Secondary Research Questions

<!-- -->

1. Does the nerve block combination facilitate earlier postoperative mobilization?
2. Does it reduce the incidence of postoperative nausea and vomiting?
3. What is the incidence of neurological complications (sensory deficits and motor impairment)?
4. Does the intervention affect length of hospital stay?

Randomization and Allocation Procedure Randomization is conducted the day before surgery by the responsible anesthesiologist using a computer-generated randomization sequence. The anesthesiologist draws a sealed randomization envelope containing the group allocation. The envelope accompanies the patient's medical record and case report forms (CRFs ) throughout the hospital stay and is verified in the operating room by the anesthesiologist.

Anesthesia type (general anesthesia with propofol and remifentanil using TCI (Target Controlled Infusion) with Eleveld pharmacokinetic model, or spinal anesthesia with 0.5% bupivacaine) is determined by clinical indication and is independent of randomization.

Arms and Interventions All patients receive standardized multimodal analgesia preoperatively: etoricoxib, paracetamol, oxycodone, and betamethasone.

Intervention Arm: Nervus Vastus Medialis (NVM) block + Saphenous Nerve (SN) block + Anterior Femoral Cutaneous Nerve (AFCN) block + Local Infilration Analgesia (LIA) All nerve blocks are performed under ultrasound guidance with strict sterile precautions.

1. NVM block:

   * In-plane ultrasound approach using a linear high-frequency transducer
   * Needle inserted from the lateral thigh, placed between vastus medialis and sartorius, lateral to the adductor membrane
   * Injection: 5 ml ropivacaine 5% with clonidine 1.875 micrograms per ml
   * NVM is visualized and surrounded by local anesthetic
2. SN block:

   - Same needle entry point as NVM block
   * Needle retracted and advanced toward the lateral border of the femoral artery
   * Sartorius posterior fascia is perforated; needle tip placed beside the SN
   * Injection: 10 ml ropivacaine 0.5% with clonidine 1.875 micrograms per ml
   * Hydrodissection of the adductor canal is observed; SN is completely surrounded by local anesthetic
3. AFCN block:

   - AFCN divides into multiple branches at the level of the femoral triangle

   - Nerves are located superficially above the superior sartorius fascia in loose subcutaneous fascia
   * Typically, 3-4 individual nerve branches are visualized
   * Needle retracted in-plane from the adductor canal approach
   * Individual branches blocked superficially above sartorius
   * Injection: 1 ml ropivacaine 5% with clonidine 1.875 micrograms per ml per branch
4. LIA:

   - LIA is administered by the surgeon before wound closure

   - 150 ml ropivacaine 2 mg/ml with 0.5 mg adrenaline is infiltrated periarticular around the knee capsule, collateral ligaments, under the patella, and subcutaneously

   Control Arm: LIA Only

   - LIA is administered by the surgeon before wound closure

   - 150 ml ropivacaine 2 mg/ml with 0.5 mg adrenaline is infiltrated periarticular around the knee capsule, collateral ligaments, under the patella, and subcutaneously

   Enrollment Planned Total Enrollment: 200 patients

   Principal Investigators:

   • Fredrik Fellert, MD, DESA, EDIC, EDEC, PhD student, Senior Consultant, VO Planned Operations, Trelleborg Hospital, Lund University, Sweden
   * Andreas Ekman, MD, PhD, DEAA, Senior Consultant, VO Planned Operations, Trelleborg Hospital, Lund University, Sweden
   * Fredrik Sjövall, MD, Associate Professor, Senior Consultant, Department of Perioperative and Intensive Care, Malmö University Hospital, Lund University, Sweden
   * Gunnar Flivik, MD, Associate Professor, Senior Consultant, Department of Orthopedics, Lund university Hospital, Lund University, Sweden

   Ethical Approval Ethics Committee: Swedish Ethical Review Authority (Etikprövningsmyndigheten) Approval Reference: 2025-06626-01 Approval Date: 2025-10-30 This study is conducted in accordance with the Declaration of Helsinki and applicable Swedish regulations for clinical research, including the Act on Ethical Review of Research Involving Humans (2003:460).

   Statistical Considerations:

   A priori sample size calculation was performed using a two-sample t test with a significance level (alpha) of 0.05 and statistical power of 0.80, assuming a between-group difference of 2 points on the NRS pain scale. This yielded an estimated requirement of 90 participants per group to achieve adequate power. Data will be analyzed using SPSS. Descriptive statistics will be presented as appropriate for the distribution of each variable. Group comparisons will be performed using chi-square test or Fisher's exact test for categorical variables, and independent-samples t test or Mann-Whitney U test for continuous variables, depending on assessment of normality.

ELIGIBILITY:
Inclusion Criteria:

-Undergoing primary unilateral total knee arthroplasty

Exclusion Criteria:

* Pregnancy
* Coagulopathy or other bleeding disorder that precludes regional anesthesia
* Allergy to local anesthetics
* Inability to understand spoken and written Swedish
* Unwillingness to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity: Measured using the NRS scale 0-10 at multiple predefined time points postoperatively (1 hour, 4 hours, 24 hours) | The day of surgery, postop day 1 and 14 days post-surgery
  Pain intensity was assessed using the Numeric Rating Scale (NRS) upon arrival at the post anesthesia care unit (PACU) and at 1, 2, 3 and 4 hours post-PACU admission, as well as at ward admission, on the evening of the surgery day, the morning of Postoperative Day 1 (POD1), and at discharge. At the post-surgery visit at 14 days NRS was also assessed.
Difference in analgesia consumption | The day of surgery, postop day 1 and 14 days post-surgery
  Total Postoperative Opioid Consumption: Cumulative morphine equivalents (mg) recorded during hospitalization (intraoperative and postoperative period).

SECONDARY OUTCOMES:
Time to mobilization | The day of surgery, postop day 1
  Time to First Mobilization: Time (hours) from arrival to the PACU to first mobilization (sitting, standing, or walking as tolerated)
Incidence of postoperative nausea and vomiting | The day of surgery, postop day 1
  Postoperative Nausea and vomiting: Incidence and severity recorded via patient report and use of antiemetic medication
Neurological complications | The day of surgery, postop day 1 and at day 14 post-surgery. Patients that report or shows neurological complications at the post surgery visit day 14 will be followed up once more, 6 month after surgery.
  Difference in frequency of neurological complications between groups: sensory deficits (paresthesia, numbness, hypoesthesia) and motor impairment (weakness, difficulty in muscular contraction) reported to and assessed by physiotherapist.
Length of Hospital Stay | 1-5 days post-surgery
  Number of postoperative days in hospital.
Difference in postoperative pain depending on method of anesthesia | The day of surgery, postop day 1 and 14 days post-surgery
  Exploratory analysis by anesthesia type: Comparison of pain scores (assessed by NRS (0-10)) and opioid consumption (equivalents in mg) between patients receiving general anesthesia versus spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ekman, MD, PhD, Principal Investigator — VO Planned Operations, Trelleborg Hospital, and Lund University, Sweden
Locations (1):
- Department of Anaesthesiology, Trelleborg Hospital, Trelleborg, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be de-identified; each patient receives a unique enrollment number. De-identified study data will be stored in an Excel spreadsheet secured behind Lund University's institutional firewall. Data will not be shared publicly. Access to anonymized datasets may be considered upon reasonable request to the principal investigators, subject to GDPR compliance and institutional review approval.
  Data Availability: Results and findings will be published in peer-reviewed journals and may be presented at scientific conferences. Individual patient data will remain confidential and protected in accordance with applicable data protection regulations.

REFERENCES:
- [Background] Bjorn S, Nielsen TD, Jensen AE, Jessen C, Kolsen-Petersen JA, Moriggl B, Hoermann R, Nyengaard JR, Bendtsen TF. The anterior branch of the medial femoral cutaneous nerve innervates the anterior knee: a randomized volunteer trial. Minerva Anestesiol. 2023 Jul-Aug;89(7-8):643-652. doi: 10.23736/S0375-9393.22.16910-5. Epub 2023 Feb 27. PMID 36852567
- [Background] Riegler G, Pivec C, Jengojan S, Mayer JA, Schellen C, Trattnig S, Bodner G. Cutaneous nerve fields of the anteromedial lower limb-Determination with selective ultrasound-guided nerve blockade. Clin Anat. 2021 Jan;34(1):11-18. doi: 10.1002/ca.23582. Epub 2020 Feb 29. PMID 32065687
- [Background] Luo ZY, Yu QP, Zeng WN, Xiao Q, Chen X, Wang HY, Zhou Z. Adductor canal block combined with local infiltration analgesia with morphine and betamethasone show superior analgesic effect than local infiltration analgesia alone for total knee arthroplasty: a prospective randomized controlled trial. BMC Musculoskelet Disord. 2022 May 19;23(1):468. doi: 10.1186/s12891-022-05388-5. PMID 35590308
- [Background] Mingdeng X, Yuzhang A, Xiaoxiao X, Yucheng A, Xin W, Dianming J. Combined application of adductor canal block and local infiltration anesthesia in primary total knee arthroplasty: an updated meta-analysis of randomized controlled trials. Arch Orthop Trauma Surg. 2022 Jun;142(6):913-926. doi: 10.1007/s00402-020-03706-x. Epub 2021 Jan 8. PMID 33417022
- [Background] Schnabel A, Reichl SU, Weibel S, Zahn PK, Kranke P, Pogatzki-Zahn E, Meyer-Friessem CH. Adductor canal blocks for postoperative pain treatment in adults undergoing knee surgery. Cochrane Database Syst Rev. 2019 Oct 26;2019(10):CD012262. doi: 10.1002/14651858.CD012262.pub2. PMID 31684698
- [Background] Berikashvili LB, Yadgarov MY, Kuzovlev AN, Smirnova AV, Kadantseva KK, Kuznetsov IV, Polyakov PA, Likhvantsev VV. Adductor Canal Block Versus Femoral Nerve Block in Total Knee Arthroplasty: Network Meta-Analysis. Clin J Pain. 2024 Jul 1;40(7):447-457. doi: 10.1097/AJP.0000000000001214. PMID 38561898
- [Background] Hasabo EA, Assar A, Mahmoud MM, Abdalrahman HA, Ibrahim EA, Hasanin MA, Emam AK, AbdelQadir YH, AbdelAzim AA, Ali AS. Adductor canal block versus femoral nerve block for pain control after total knee arthroplasty: A systematic review and Meta-analysis. Medicine (Baltimore). 2022 Aug 26;101(34):e30110. doi: 10.1097/MD.0000000000030110. PMID 36042669
- [Background] Wang D, Yang Y, Li Q, Tang SL, Zeng WN, Xu J, Xie TH, Pei FX, Yang L, Li LL, Zhou ZK. Adductor canal block versus femoral nerve block for total knee arthroplasty: a meta-analysis of randomized controlled trials. Sci Rep. 2017 Jan 12;7:40721. doi: 10.1038/srep40721. PMID 28079176
- [Background] Peng XQ, Fei ZG, Sun CG, Zhou QJ. Efficacy and safety of local infiltration analgesia for pain management in total knee and hip arthroplasty: A meta-analysis of randomized controlled trial. Medicine (Baltimore). 2020 May 29;99(22):e20640. doi: 10.1097/MD.0000000000020640. PMID 32481477
- [Background] Marques EM, Jones HE, Elvers KT, Pyke M, Blom AW, Beswick AD. Local anaesthetic infiltration for peri-operative pain control in total hip and knee replacement: systematic review and meta-analyses of short- and long-term effectiveness. BMC Musculoskelet Disord. 2014 Jul 5;15:220. doi: 10.1186/1471-2474-15-220. PMID 24996539